CLINICAL TRIAL: NCT03295578
Title: Blood Glucose Monitoring, Cognition, and Wellbeing in Relation to Food Intake @ Work - a Pilot Study
Brief Title: Blood Glucose, Cognition and Wellbeing @ Work
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TNO (Other)
Collaborators: Wageningen University and Research (Other); Jumbo Supermarkten Bv. (Unknown); Noldus Information Technology B.V. (Unknown); Google LLC. (Industry)
Responsible Party: Principal Investigator, Iris de Hoogh, Research Scientist, TNO
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: P9663
Record Dates: First submitted 2017-09-12; First posted 2017-09-28 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Healthy; PreDiabetes
Keywords: employees; continuous glucose monitoring; personalized feedback; cognition; wellbeing
MeSH Terms: conditions — Prediabetic State | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with two parallel arms.
Who Masked: Participant, Investigator
Masking Description: Participants will be assigned to the personalised feedback group or generic feedback group (control) by an independent researcher that is not involved in the study. Assignment will be random and balanced for gender and age. To avoid subjects being aware of the group they are in, both groups will receive some sort of feedback, either generic or personalised. Subjects will be informed that they should not discuss their feedback with other study participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Personalized feedback group (Experimental): In between the two measurement periods, the personalized feedback group will receive an explanation and personalized feedback on their self-measured data (interstitial glucose, cognition, wellbeing and food intake).
  Interventions: Other: Personalized feedback; Device: Continuous glucose monitoring device
- General feedback group (Placebo Comparator): The generic feedback group will receive a generic explanation about glucose, cognition wellbeing and food intake and their relationship. The generic feedback will not include personal results.
  Interventions: Other: Generic feedback; Device: Continuous glucose monitoring device

INTERVENTIONS:
Other: Personalized feedback — The personalized feedback report will contain a general explanation about glucose, cognition and wellbeing, healthy cut-offs and/or benchmark values, and why these measures are relevant for personal health and wellbeing. Also, a general explanation will be given about how glucose levels can be influenced.
  Also, the personalized feedback will contain the individual glucose response profiles, as well as graphs showing the wellbeing scores over time. The registered food intake will be mapped and linked to the glucose and wellbeing profiles. The results of the wellbeing questionnaire will also be shown and will be linked to the individual profiles and food intake.
  Other Names: personalized feedback report
  Arms: Personalized feedback group
Other: Generic feedback — The generic feedback will contain a generic explanation about glucose, cognition wellbeing and food intake and their relationship. The generic feedback will not include personal results.
  Other Names: Generic feedback report
  Arms: General feedback group
Device: Continuous glucose monitoring device — This is not an intervention, but a measurement device used during the study. Added here as intervention to avoid errors in the system.
  Other Names: Abbott FreeStyle Libre Pro

SUMMARY:
This randomized controlled pilot study has as a main aim to investigate the relationship between glucose and cognition and wellbeing, as well as food intake in an at-work setting. Additionally, the continuous glucose data collected in the study will be used to investigate the inter- and intraindividual variability in glucose response to foods/meal in a real-life setting.

Finally, the study aims to determine if self-monitoring and feedback about food intake and health stimulate individuals to make healthier choices.

This study will have two groups, the feedback group and the control group. The study will consist of two self-monitoring periods of two weeks. In between these two self-monitoring periods, the participants in the feedback group will be given feedback on their measurement data. The control group will not get any feedback.

DETAILED DESCRIPTION:
Many people in the Western world have an unhealthy lifestyle, including an unhealthy dietary pattern. Numerous approaches have been taken to stimulate people to maintain a more healthy diet, but results are highly variable across studies and subjects. One explanation for this is that in many approaches the individuals' specific needs and the context they live and work in are not sufficiently taken into account. For an approach to be more effective, personal characteristics need to be taken into account. In other words, the approach needs to be tailored or personalised. When focussing on personalized nutrition and health in the work environment, the aspects of health that are included in the study should also be relevant for the work environment. Three main parameters of interest are selected: (postprandial) blood glucose levels, cognition and (subjective) wellbeing.

Objective:

The primary objective of this pilot study is to investigate the relationship between glucose and cognition and wellbeing, as well as food intake in an at-work setting.

Secondary objectives are :1) Does self-monitoring and feedback about food intake and health stimulate individuals to make healthier choices? 2) What are the user experiences of employees to perform self-monitoring of and receive feedback on, glucose, wellbeing and cognition in the workplace?

Study design:

This study will be designed as a randomized controlled trial with two groups, the feedback group and the control group. The study will consist of two self-monitoring periods of two weeks. In between these two self-monitoring periods, the participants in the feedback group will be given feedback on their measurement data. The control group will not get any feedback.

Study population:

Forty participants, both men and women, will be recruited from the staff at the head-quarters of Jumbo supermarkets in Veghel. Inclusion criteria are presence at head-quarters for at least 4 days per week and frequent visitors of the company lunch restaurant. Exclusion criteria are shift work, diabetic patients, neurological or psychiatric complaints and specific food-related allergies.

Intervention:

The intervention consists of standardized meals and personalized feedback. During the first two-week measurement period study participants will be asked to consume standardized lunches at work days in the company restaurant. In between the two measurement periods, the feedback group will receive personalized feedback on their self-measured data (interstitial glucose, cognition, wellbeing, and food intake). At the end of the second measurement period both the feedback group and the control group will receive a personalized feedback form, including a debriefing about the study.

Main study parameters/endpoints:

Primary endpoints are self-monitored daily food intake, glucose levels, cognitive performance, and wellbeing.

ELIGIBILITY:
Inclusion Criteria:

* Must be present at Jumbo head-quarters during lunch at least four days/week and have access to their computer for one hour after lunch during the two 2-week self-monitoring periods
* Must be frequent visitors of the company lunch restaurant (Jumbo food café), with a minimum of three times per week
* Having giving written informed consent
* Willing to comply with all study procedures

Exclusion Criteria:

* Shift workers
* Diabetes type 2 patients
* Under treatment for neurological or psychiatric complaints, including eating disorders
* Specific dietary preferences, including vegan, raw food, paleo. Vegetarian, pescetarians and flexitarians can participate in the study
* Allergies or intolerances, including coeliac disease, gluten intolerance, lactose intolerance, milk protein allergy
* Skin allergy or eczema

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2017-11-17 (Actual); Study Completion 2017-12-22 (Actual)

PRIMARY OUTCOMES:
Daily glucose levels | Continous (sampled every 15 minutes for a duration of 14 days)
  measured using a continuous glucose monitoring device
Daily food intake | daily registration of food intake during working hours for a duration of 14 days (during both the two week measurement periods)..
  measured using a food intake application
Cognition tests | twice per day (before and after lunch) at working days for a duration of 14 days, during both the two week measurement periods
  via Smartphone application. Tests include direct recall, free recall & delayed recall.
Wellbeing | This questionnaire will be administered five times per day; two times in the morning, once five minutes before lunch (before with cognition test), once one hour after lunch (before cognition test) and once in the afternoon for two times 14 days.
  via Smartphone application. Includes VAS scales for including five questions for 'feeling energetic - tired, 'feeling focused - distracted', 'feeling positive - negative' , 'feeling motivated - unmotivated' , 'feeling relaxed - stressed'

SECONDARY OUTCOMES:
Intention to eat healthy | baseline and after eight weeks (end of study)
  measured with three items on seven-point scales from totally disagree (1) to totally agree (7). The items are 'I'm planning on eating healthy', 'I would consider to eat healthy' and 'I'm absolutely going to eat healthy'.
Quantitative user experiences | baseline and after eight weeks (end of study)
  Self-efficacy towards maintaining a healthy diet and type of motivation to eat healthy
Qualitative user experiences | four short surveys (baseline, day 1, after two weeks, after eight weeks) and in focus groups after eight weeks
  the survey includes self-constructed scales that measure user experience with the research in general, self-monitoring devices and personal feedback. Focus groups are needed to understand the reasoning behind the answers that employees give in the surveys and to validate initial analysis of the survey.

OTHER OUTCOMES:
Focus on future consequences | baseline
  validated questionnaire from Joireman et al (2012). Output will be used as input for formulating the personalized feedback
Subjective health | Baseline and after eight weeks (end of study)
  • Subjective health is measured with two items that are rated on seven-point scales from 'very unhealthy' (1) to 'very healthy' (7).
Eating habits (at the workplace) | Baseline and after eight weeks (end of study)
  mapped via a questionnaire, concerning how often one eats breakfast and snacks, how often one eats in the company restaurant at work, how often one brings their own lunch or buys their lunch, how often one goes on lunch walks etc.
Physical activity | Baseline and after eight weeks (end of study)
  the Dutch Norm for Healthy Physical Activity.
BMI | Baseline and after eight weeks (end of study)
  calculated based on self-reported height and weight

CONTACTS AND LOCATIONS:
Overall Officials: Iris M de Hoogh, Msc, Principal Investigator — TNO (Netherlands Organization for Applied Scientific Research)
Locations (1):
- Jumbo Supermarkten BV., Veghel, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: No